CLINICAL TRIAL: NCT02545790
Title: Cardiac Remodeling and Circulating Biomarkers in Pediatric Left Ventricular Pressure Loading Lesions
Acronym: LVOTO
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 15-0635
Record Dates: First submitted 2015-09-02; First posted 2015-09-10 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Coarctation of Aorta; Aortic Stenosis; Cardiac Hypertrophy
Keywords: coarctation of aorta; aortic stenosis; biomarkers; cardiac hypertrophy
MeSH Terms: conditions — Aortic Coarctation; Aortic Valve Stenosis; Cardiomegaly

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and tissue samples from patients will be stored for the duration of the study. Patients may choose to consent to have these samples stores beyond the completion of primary analysis for testing in future studies.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Persistent hypertrophy: Elevated cardiac mass at follow-up time point as measured by Echocardiographic and Serologic evaluations.
  Interventions: Procedure: Echocardiogram; Biological: Serology
- Normal geometry: Normal cardiac mass at follow-up time point as measured by Echocardiographic and Serologic evaluations.
  Interventions: Procedure: Echocardiogram; Biological: Serology

INTERVENTIONS:
Procedure: Echocardiogram — 2 and 3-dimensional echocardiographic images will be obtained to estimate LV mass, ejection fraction (Simpson's biplane), fractional shortening (M mode Doppler), and pulse-wave estimated pressure gradient across the outflow obstruction.
  Other Names: Diagnostics
Biological: Serology — protein analysis targeting several potential protein biomarkers for cardiac remodeling and hypertrophy as well as targeting known miRNAs.
  Other Names: Diagnostics

SUMMARY:
This study is designed to learn more about children who have blockage of the left side of their heart. The goal is to determine how much the heart muscle has thickened before surgery and how it changes in the months after surgery. Investigators are also looking for blood tests that may help them predict which patients will have the most thickening pre-operatively and the best return towards normal after surgery. The findings of this study will help the investigators develop new tests to monitor affected patients and develop new therapies to help minimize heart thickening.

ELIGIBILITY:
Inclusion Criteria:

* Congenital heart disease patients with the following diagnoses undergoing surgical repair: Coarctation of the aorta (CoA), aortic stenosis (AS), subaortic membrane (sub-AS), supravalvar aortic stenosis (supra-AS).
* All patients will have age from birth through 18 years of age.
* While we will generally not enroll patients with other co-morbid heart disease that would alter the cardiac physiology (see exclusion criteria), patients with patent foramen ovale, atrial septal defect, and patent ductus arteriosus specifically will be allowed.

Exclusion Criteria:

* Patients with lesions not listed in inclusion criteria (including but not limited to hypoplastic left heart syndrome, Shone's complex, mitral valve stenosis or regurgitation greater than trivial, non-restrictive ventricular septal defect, interrupted aortic arch, atrio-ventricular canal defect)
* Corrected gestational age at time of surgery <34 weeks
* Weight at time of surgery <2000g.
* Patients who will not be seen for any follow-up care at Children's Hospital Colorado

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Potential subjects will be identified from the cardiac surgical and clinic schedules at Children's Hospital Colorado (CHCO).
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Left ventricular mass | 1 year after surgery
  Left ventricular mass will be measured by 2D echocardiography at 1 year after surgical correction.
Change in left ventricular mass | Within 1 week prior to surgery, 24-72 hrs after surgery, 1 year after surgery
  Left ventricular mass will be measured by 2D echocardiography prior to surgery, immediately after surgery, and will be compared to that measured at 1 year after surgical correction.

SECONDARY OUTCOMES:
Relative wall thickness | 1 year after surgery
  A more detailed measure of relative wall thickness (RWT) will be assessed by echocardiography at 1 year after surgical correction.
Left ventricular mass | 1 year after surgery
  Left ventricular mass will be measured by 3D echocardiography at 1 year after surgical correction.
Change in relative wall thickness | Within 1 week prior to surgery and 1 year after surgery
  Relative wall thickness will be measured by 2D echocardiography prior to surgery and at 1 year after surgical correction.
Change in relative wall thickness | 24-72 hours and 1 year after surgery
  Relative wall thickness will be measured by 2D echocardiography 24-72 hours and at 1 year after surgical correction.
Change in left ventricular mass | 24-72 hours and 1 year after surgery
  Change in left ventricular mass will be measured by 3D echocardiography 24-72 hours and 1 year after surgical correction.
Change in left ventricular mass | Within 1 week prior to surgery and 1 year after surgery
  Change in left ventricular mass will be measured by 3D echocardiography prior to surgery and at 1 year after surgical correction.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin S Frank, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Denver, Colorado, United States